CLINICAL TRIAL: NCT02084875
Title: A Phase 1, Randomized, Open Label, Single Dose, 2-Period Crossover Study To Evaluate The Effect Of Food On The Pharmacokinetics Of Tofacitinib Modified Release (MR) 11 Mg Tablets In Healthy Western And Japanese Volunteers
Brief Title: A Study To Evaluate The Effect Of Food On The Behavior Of Tofacitinib Modified Release 11 Milligram Tablets In Healthy Western And Japanese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A3921180
Record Dates: First submitted 2014-03-10; First posted 2014-03-12 (Estimated); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Healthy
Keywords: Food effect; pharmacokinetic; healthy volunteer
MeSH Terms: interventions — Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- tofacitinib MR 11 mg Fed (Experimental): tofacitinib modified release (MR) 11 mg tablet administered with food.
  Interventions: Drug: tofacitinib modified-release (MR) formulation
- tofacitinib MR 11 mg Fasting (Experimental): tofacitinib modified release (MR) 11 mg tablet administered without food.
  Interventions: Drug: tofacitinib modified-release (MR) formulation

INTERVENTIONS:
Drug: tofacitinib modified-release (MR) formulation — A single dose of tofacitinib modified release 11 mg tablet after receiving the standard FDA high fat/high calorie meal.
  Arms: tofacitinib MR 11 mg Fed
Drug: tofacitinib modified-release (MR) formulation — tofacitinib modified release (MR) 11 mg tablet after a 10 hour overnight fast.
  Arms: tofacitinib MR 11 mg Fasting

SUMMARY:
This study will evaluate the drug behavior and safety of a single dose of the 11 milligram tofacitinib (CP-690,550) modified-release formulation in 24 healthy volunteers when taken after eating a high fat meal (the effect of food). This will be compared to the drug behavior and safety of a single dose of the 11 milligram tofacitinib (CP-690,550) modified-release formulation when taken after a 10 hour fast.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers and/or healthy females volunteers of non-childbearing potential who are 18 to 55 years of age;
* Healthy volunteers who are of Japanese or Western descent;
* Healthy volunteers with no evidence of active or latent or inadequately treated tuberculosis.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease;
* Clinically significant infections within the past 3 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-04-11 (Actual); Primary Completion 2014-05-25 (Actual); Study Completion 2014-05-25 (Actual)

PRIMARY OUTCOMES:
Area under the curve from time zero to infinity | 48 hours post dose
  Area under the curve from time zero to infinity
Area under the plasma concentration-time profile from time zero to time of the last quantifiable concentration | 48 hours post dose
  Area under the plasma concentration-time profile from time zero to time of the last quantifiable concentration
Maximum Observed Plasma Concentration (Cmax) | 48 hours post dose
  Maximum Observed Plasma Concentration (Cmax)

SECONDARY OUTCOMES:
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 48 hours post dose
  Time to peak concentration
Plasma Decay Half-Life (t1/2) | 48 hours post dose
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Glendale Adventist Medical Center, Glendale, California, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921180&StudyName=A%20Phase%201%2C%20Randomized%2C%20Open%20Label%2C%20Single%20Dose%2C%202-period%20Crossover%20Study%20To%20Evaluate%20The%20Effect%20Of%20Food%20On%20The%20Pharmacokinetics%20Of%20Tofacitinib%20Modified%20Release%20%28mr%29%2011%20Mg%20Tablets%20In%20Healthy%20Western%20And%20Japanese%20Volunteers